CLINICAL TRIAL: NCT00704054
Title: A Multi-Center Phase I Study of Intravenous Deforolimus (AP23573, MK-8669) Administered QDX5 Every Other Week in Pediatric Patients With Advanced Solid Tumors
Brief Title: A Multi-Center Phase I Study of Intravenous Deforolimus (AP23573, MK-8669) Administered QDX5 Every Other Week in Pediatric Patients With Advanced Solid Tumors (8669-028)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); Pediatric Cancer Foundation (Other); University of Colorado, Denver (Other); Johns Hopkins All Children's Hospital (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-028; SUN08-01 (Other Grant/Funding Number: SUN08-01 Pediatric Cancer Foundation); AP23573-07-110
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Solid Tumors
Keywords: Pediatric; Solid Tumor; CNS Tumor; Lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma | interventions — ridaforolimus

ARMS (1):
- 1 (Experimental): Ridaforolimus is given as an IV infusion over 30 minutes on days 1-5 and 15-19 of each 28 day cycle. For children less than 10 kg body weight, dosing will be adjusted.
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — Ridaforolimus is given as an IV infusion over 30 minutes on days 1-5 and 15-19 of each 28 day cycle. For children less than 10 kg body weight, dosing will be adjusted.
  Other Names: AP23573, deforolimus, MK-8669

SUMMARY:
Ridaforolimus (Deforolimus, AP23573, MK-8669) is an mTor inhibitor shown to have promising activity in adults with a variety of solid malignancies, particularly the sarcomas. To date, no studies to evaluate appropriate dosing or to obtain pharmacokinetic data in pediatric patients have been conducted. Sarcomas are the second most common solid malignancies in children and young adults, and for those patients with recurrent or refractory disease, new therapies are needed. This initial evaluation of ridaforolimus will help define appropriate dosing and toxicity evaluations, as well as establish the first pharmacokinetic and biologic correlative data in pediatric patients treated with ridaforolimus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 1 to <18 years at the time of study entry for the dose escalation portion of the study
* Histologic diagnosis of a malignant lymphoma or solid tumor, including tumors of the central nervous system that has progressed in the opinion of the investigator despite standard therapy or for which no effective standard therapy is known
* Patients may have measurable or non-measurable disease as defined by RECIST
* Patients with brainstem glioma or intrinsic pontine glioma do not need biopsy proof of the diagnosis, but must have documentation at their local institution that there is agreement among the attending oncologist and/or neuro-oncologist, radiologist, and neurosurgeon/pediatric neurosurgeon that the diagnostic imaging studies are consistent with a diagnosis of brainstem or intrinsic pontine glioma
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, surgery or radiotherapy prior to entering this study
* Performance Status: EGOG 0-2 for patients age 16 and older; Karnofsky >40% for patients >10 years of age; Lansky Play Scale >40 for children < 10 years of age
* Life expectancy greater than or equal to 12 weeks
* There is no limit to the number of prior treatment regimens provided that performance status, organ function, and life expectancy meet the study criteria
* No persistent toxicities from previous therapies > Grade 2 by NCI CTCAE version 3. For patients with CNS tumors ONLY, if baseline neurotoxicity due to primary tumor involvement or post-operative complications, Grade 3 neurotoxicity is allowed if stable
* Normal organ and marrow function
* For females of childbearing potential, a negative pregnancy test must be documented prior to enrollment
* Patients who enter this study and their sexual partners who are of childbearing potential must agree to use an effective form of contraception

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within three (3) weeks (or six weeks for nitrosoureas or mitomycin C) prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients receiving any other investigational agents or using any investigational devices
* Patients with leukemia
* Patients who have previously received deforolimus or other rapamycin analogs
* History of allergic reactions (in opinion of the investigator) attributed to compounds of similar chemical or biologic composition to deforolimus and its excipients used in administration
* Uncontrolled intercurrent illness
* Pregnant women are excluded from this study because the teratogenic or abortifacient effects of deforolimus are not known at this time
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, known HIV-positive patients are excluded from the study because of possible pharmacokinetic interactions with deforolimus
* Autologous or allogeneic stem cell transplant <3 months prior to enrollment; any evidence of on-going graft versus host disease (GVHD), or GVHD requiring immunosuppressive therapy. Patients who have had prior stem cell transplant regimens must be discussed with and approved by the principal investigator prior to registration

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To establish the DLT and the MTD of ridaforolimus administered daily x 5 every 14 days in pediatric patients with recurrent/refractory solid tumors, including lymphoma and tumors of the central nervous system. | Duration of trial

SECONDARY OUTCOMES:
To determine the pharmacokinetic and pharmacodynamic properties of ridaforolimus in pediatric patients with recurrent/refractory solid tumors, including tumors of the central nervous system. Screening at Day 1-18, Cycle 2 Day 1, Cycle 2 Day 15. | Duration of trial
To evaluate the safety and efficacy data of ridaforolimus when administered at the MTD or recommended phase II dose and schedule in an expanded cohort of patients when administered daily x 5 every 14 days | Duration of trial
To assess pharmacogenomic parameters from archival tumor specimens that may correlate with response to ridaforolimus. | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Gore, MD, Principal Investigator — University of Colorado, Denver; Christopher Turner, MD, Study Director — Ariad Pharmaceuticals

REFERENCES:
- [Result] Gore L, Trippett TM, Katzenstein HM, Boklan J, Narendran A, Smith A, Macy ME, Rolla K; Pediatric Oncology Experimental Therapeutics Investigators' Consortium (POETIC); Narashimhan N, Squillace RM, Turner CD, Haluska FG, Nieder M. A multicenter, first-in-pediatrics, phase 1, pharmacokinetic and pharmacodynamic study of ridaforolimus in patients with refractory solid tumors. Clin Cancer Res. 2013 Jul 1;19(13):3649-58. doi: 10.1158/1078-0432.CCR-12-3166. Epub 2013 May 9. PMID 23659969
- See also: Pediatric Cancer Foundation — http://www.pcfweb.org/